CLINICAL TRIAL: NCT06699745
Title: Comparison of the Effects of Music and White Noise on Fear, Anxiety and Pain Levels in Children Performed Endoscopy
Brief Title: Comparison of the Effects of Music and White Noise in Children Performed Endoscopy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Busra Inac Yilmaz, IstanbulUC, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IUC-LEE-BIY-26
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: School Age Children; Endoscopy, Gastrointestinal
Keywords: endoscopy; fear; anxiety; pain; music; white noise
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- white noise group (Experimental): Children in the group will be made to listen to white noise at an appropriate decibel level.
  Interventions: Behavioral: white noise intervention
- music group (Experimental): Music will be listened at an appropriate decibel level for the children in the group.
  Interventions: Behavioral: Music intervention
- control group (No Intervention): No application was made to the control group.

INTERVENTIONS:
Behavioral: Music intervention — In studies, white noise was used as a sedative in infants. It was not used in older children. In school-age children, white noise will be used to reduce fear, anxiety and pain during the endoscopy procedure.
  Arms: music group
Behavioral: white noise intervention — White noise will be played at a decibel level appropriate for the children in the group.
  Arms: white noise group

SUMMARY:
The study was planned as a randomized controlled experimental study to compare the effects of music and white noise on fear, anxiety and pain levels before, during and after the procedure in school-age children (6-12 years old) who will undergo endoscopy.

Hypothesis 0 (H0): There is no difference in fear, anxiety, pain, parental anxiety and pulse, respiration and oxygen saturation values between children exposed to music and white noise.

Hypothesis 1 (H1): Children who were exposed to music and white noise had lower fear scores than children who were not exposed to any application.

Hypothesis 2 (H2): Children who were exposed to music and white noise had lower anxiety scores than children who were not exposed to any application.

Hypothesis 3 (H3): Children who were exposed to music and white noise had lower pain scores than children who were not exposed to any application.

Hypothesis 4 (H4): Children who were exposed to music and white noise had lower pulse value scores than children who were not exposed to any application.

Hypothesis 5 (H5): Children who were exposed to music and white noise had lower respiratory rate scores than children who were not exposed to any application.

Hypothesis 6 (H6): Children who were exposed to music and white noise had higher oxygen saturation value scores than children who were not exposed to any application.

Hypothesis 7 (H7): Parents of children who were exposed to music and white noise had lower parental anxiety than parents of children who were not exposed to any treatment.

There are music group, white noise and control group in the study.

DETAILED DESCRIPTION:
The independent variables of the study are age, gender, music and white noise application.

The dependent variables are; Children's Fear Scale (CFS) scores used to measure children's fear, Children's Anxiety Scale-State (CAS-D) scores used to measure anxiety, The Faces Pain Scale Revised (FPS-R) scores used to measure pain status, pulse, respiratory rate and oxygen saturation values and Beck Anxiety Inventory scores obtained from parents.

ELIGIBILITY:
Inclusion Criteria:

* School age (6-12 years old) child,
* Have not had an endoscopy procedure before,
* Have not had a surgical procedure before,
* Have been requested to have an endoscopy by a physician,
* Be able to communicate,
* Have no hearing or speech problems,
* Agree to participate in the study,
* Have not used analgesics for 6 hours before the procedure,
* The child can count from 1 to 10,
* Have the ability to order numbers (knowing that numbers are big or small (e.g. 6 is less than 7, 4 is greater than 2, etc.).

Exclusion Criteria:

* Not being of school age (under 6 years old, over 12 years old),
* Having had an endoscopy procedure before,
* Having had a surgical procedure before,
* Not being able to communicate,
* Having hearing and speech problems,
* Not agreeing to participate in the study,
* Having used analgesics up to 6 hours before the procedure,
* The child not having the ability to sort and count numbers.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Child fear scale | six months
  The Child Fear Scale (CFS), developed by McMurty and colleagues (2011), consists of five drawn facial expressions ranging from a neutral expression (0 = no anxiety) to a frightened face (4 = severe anxiety). The validity and reliability of the scale were performed by Gerçeker and colleagues (2018). The CGI value for the CFS is 0.89 (McMurty et al., 2011).
Child anxiety scale-state | six months
  The Child Anxiety Scale State (CAS-S) developed by Ersig et al. (2013) is used to measure the anxiety of the child's current situation. The validity and reliability of the scale were made by Gerceker et al. (2018). The Content Validity Index (CVI) value for CAS-S was found to be 1.00.
The Faces Pain Scale - Revised | six months
  It is a self-report measure of pain intensity developed for children. It has been made more suitable for use by using visual depictions of six facial expressions representing increasing levels of pain intensity and by adapting the metric scoring to 0-10. The revised version of the facial pain scale is widely used in the adult and pediatric populations for pain intensity assessment. It is easy to apply and does not require any equipment other than the faces in the picture.

SECONDARY OUTCOMES:
Beck Anxiety Inventory | six months
  Developed by Beck et al. (1988). The Cronbach alpha coefficient of the original scale is .93. The Turkish adaptation of the Beck Anxiety Inventory was prepared by Ulusoy et al. (1998). In the Turkish validity and reliability study of the scale, Cronbach alpha coefficient was determined as .93. The Beck Anxiety Inventory is a 21-question scale that individuals can answer on their own. Questions are scored between 0 and 3. The minimum score is 0 and the maximum score is 63. The total score is used in the evaluation of the scale. Increasing scores on the scale indicate an increase in the anxiety level.
pulse value | six months
  In the study, the child's pulse value was measured from the calibrated monitor before, during and after the endoscopy procedure.
respiratory value | six months
  In the study, the child's respiratory value was measured from the calibrated monitor before, during and after the endoscopy procedure.
oxygen saturation value | six months
  In the study, the child's respiratory value was measured from the calibrated monitor before, during and after the endoscopy procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Busra Inac Yilmaz, MD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Avcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I think it is not appropriate to share all information in terms of patient privacy.